



# XIENCE Xpediton Everolimus-Eluting Coronary Stent Post Marketing Surveillance

Protocol number: 14-306

**Execution Overview** 

[2.25 mm diameter stent]

# Abbott Vascular Japan Co., Ltd.

The Ministry of Health, Welfare and Labor requires this post-marketing surveillance as a condition of XIENCE Xpedition Everolimus-Eluting Coronary Stent System approval for 2.25mm stent. Your kind cooperation in this surveillance will be highly appreciated.

< This is a translation of the Japanese Version Created on: 5/29/2014 Ver. 1.0>



14-306 Version 1.0 

Approval Number 22500BZX00309000

Approval Date May 20, 2014

Generic Name of the Device Coronary Stent

Brand Name of the Device XIENCE Xpedition Everolimus-Eluting Coronary

Stent

2.25mm stent

Surveillance Period July 01, 2014 – March 31, 2021

Sponsor Abbott Vascular Japan Co., Ltd.

3-5-27 Mita, Minato-ku, Tokyo 108-6304

Responsible Manager for Post- Noriyuki Niki

marketing Surveillance Post-marketing surveillance group,

Clinical Research

Abbott Vascular Japan Co., Ltd.

#### 1. PURPOSE OF THIS SURVEILLANCE

This post-marketing surveillance (hereinafter referred to as "the PMS") is to be conducted for a medical device prescribed in Paragraph 1 in Article 14 of the Pharmaceutical Affairs Law (Law No. 145, August 10, 1960, hereinafter referred to as "PAL") by a marketing approval holder or restrictive foreign approval holder of medical device prescribed in the standard for post-marketing surveillance and post-marketing study (excluding those set forth in Ministerial Ordinance Concerning the Standards for Executing Clinical Tests on Medical Devices, Ministerial Ordinance No. 36, March 23, 2005), which is part of the standard established by the Minister of Health, Welfare and Labor set forth in Paragraph 4 in Article 14-4 and Paragraph 4 in Article 14-6 (including when applied mutatis mutandis to Paragraph 4 in Article 19 of PAL). The objectives of the PMS are to observe the frequency, type, and degree of device deficiency to assure the safety of the new medical device as well as to collect information on evaluation of the efficacy and safety for reevaluation.

The PMS is to be conducted in accordance with Ministerial Ordinance Concerning the Standards for Post-marketing Surveillance and Tests of Medical Devices (Ministerial Ordinance No. 36, March 23, 2005, hereinafter referred to as "Good Post-marketing Study Practice: GPSP").

#### 2. ELIGIBILITY AND PLANNED REGISTRATION

#### 2.1 Target Patient Population

Based on GPSP regulation, general patient population with ischemic heart disease who are eligible for treatment with XIENCE Xpedition Everolimus-Eluting 2.25mm Stent (Approval Number: 22500BZX00309000; Approval Date: May 20, 2014), will be registered, with no particular inclusion/exclusion criteria, and may be eligible for angiographic follow-up at eight months and clinical follow-up at one year.

#### 2.2 Enrollment Method

- In cases where patient informed consent (or providing some type of information) is required for PMS per the participating site policy, the Sponsor will cooperate as needed.
- If it is known at the time of index procedure that the patient is not able to return for the 8-month follow-up visit for angiogram and for the 1-year clinical follow-up, then the patient should not be registered in the PMS.
- Patients who are attending or will attend other PMS with invasive medical procedure will not be registered.
- Patients who are treated by XIENCE Xpedition 2.25mm stent will be registered.
  - The observations will be compiled on a per-patient basis even if multiple XIENCE Xpedition 2.25mm stents are implanted during the index procedure.



- A patient whose side-branch is treated by XIENCE Xpedition 2.25mm stent can be registered. In such a case, main vessel should be treated by XIENCE Xpedition.
- The observations will not be compiled on a per-patient basis if a patient is treated by XIENCE Xpedition 2.25mm stent overlapped with other stents for bail-out purpose.
- Additional revascularization procedures as a part of AE treatment and planned staged procedures will not be considered as another registration, or adverse events.
- A patient who is treated, but failed to be implanted by XIENCE Xpedition 2.25mm stent and finally treated by other devices only (No XIENCE Xpedition 2.25mm stent are implanted) must also be registered. In such a case, only the stent information, device deficiency information and reportable adverse events related to the Xpedition stent, if any, are required to be captured. Follow-up of the patient who does not receive any XIENCE Xpedition 2.25mm stent is not required.
- A patient may have another lesion(s) that may be treated by larger diameter (≥ 2.5mm) stent(s). In such a case, treatment by XIENCE Xpedition is preferable. Lesion(s) treated by other than XIENCE Xpedition 2.25mm stent is not considered as the target lesion.

# 2.3 Number of Patients to be Registered

The goal is to register about 100 patients from approximately 10 sites.

The XIENCE Xpedition 2.25 mm stent is identical to the stent of the XIENCE PRIME SV Everolimus-Eluting Coronary Stent System (Approval No. 22500BZX00070000) which is currently under use result surveillance. The sample size is calculated based on the following statistical hypothesis and assumptions: The in-stent late loss = 0.2 mm (SD = 0.5 mm) for both the XIENCE PRIME SV stent and the XIENCE Xpedition 2.25 mm stent; the QCA follow-up rate of the XIENCE PRIME SV PMS (300 patients) = 75% (225 lesions); one-tailed test with alpha = 0.05; power = 90%; non-inferiority delta = 0.195 mm. Given the above assumptions, 75 patients are needed to demonstrate the non-inferiority to the XIENCE PRIME SV stent. Assuming drop-outs, approximately 100 patients are considered a target sample size which ensures the effectiveness of the XIENCE Xpedition 2.25 mm stent.

# 3. PMS DURATION

Patients will be followed by 5 years. After signing the contract with each sites and the enrollment can be started, the target duration of patient registration for the PMS will be by September 5<sup>th</sup>, 2015.

Annual reports will be submitted to PMDA every year. After the re-submission, data will continue to be collected until 5 year follow-up is complete for all patients.

Patient data from the following time points will be collected



14-306 Version 1.0 

- Baseline (before procedure)
- Procedure
- Post-Procedure through discharge
- 8 months follow-up (follow-up angiogram)
- 1 year post-procedure (site visit is recommended)
- 2 year post-procedure (site visit/telephone contact)
- 3 year post-procedure (site visit/telephone contact)
- 4 years post-procedure (site visit/telephone contact)
- 5 years post-procedure (site visit/telephone contact)

#### 4. PATIENT TREATMENT

Patient treatment strategy should be determined by the physicians based on standard PCI procedure at each of the sites. Physicians should review the latest updated IFU, and carefully consider contraindications, warnings, and precautions when considering patient treatment.

Although dual antiplatelet management is ultimately determined by physicians, enrolled patients will be encouraged to receive adjunctive antiplatelet therapy consisting of an indefinite duration of aspirin in addition to a required minimum of 12 months of thienopyridine (clopidogrel, ticlopidine, etc.). It is recommended that physicians review the requirements of the most recent thienopyridine IFU before treating patients.

#### 5. OBSERVATION ITEMS AT EACH TIME POINT

#### **5.1** Baseline Information

#### 1) Patient Basic Information

- Index Procedure Date (Date of Registration)
- Birth year and month
- Implant of XIENCE Xpedition 2.25mm stent (Only basic information, non-implant stent form and device deficiency form must be completed in the case all XIENCE Xpedition 2.25mm stents are failed to implant)
- Gender
- Height
- Weight
- Admission and Discharge dates

# 2) Cardiac Status at the Index Procedure and Cardiac History

- Cardiac Status (Symptom of ischemia) at the Registration
- History of Myocardial Infarction
- Previous CABG
- Previous PCI

#### 3) Risk Factors

- Family History of Premature Coronary Artery Disease
- Smoking History
- Hypertension
- Dyslipidemia
- Diabetic Mellitus
- Renal Disease
- History of Stroke
- History of Major Bleeding
- Unstable Arrhythmia
- Chronic Anticoagulant Therapy

# 4) Pre-Procedure ECG

### 5) Pre-Procedure Cardiac Enzyme and Creatinine

- Cardiac Enzyme
  - o CK
  - o CK-MB (If MI is suspected then must be measured per site standard practice)
- Serum Creatinine

#### 6) Pre-Procedure Antiplatelet

- Aspirin
- Clopidogrel
- Ticlopidine
- Cilostazol

#### **5.2** Procedure Information

# 1) General Information

- Physician Name
- Procedure Start Time (Insertion of Guide Catheter)
- Procedure End Time (Removal of Guide Catheter)
- Access Site
- Number of Diseased Vessels
- Number of Treated Lesions
  - o Treated only by XIENCE PRIME (Target Lesion)
  - Treated by XIENCE PRIME and Other Stent (Target Lesion)
  - o Treated only by other devices (Non-target Lesion)
- LVEF

# 2) Lesion Information

Angiographic corelab analysis data will be adopted when it is applicable.

- Lesion Number
- Target or Non-target Lesion
- AHS Lesion Segment Number
- Lesion Type (de novo or restenosis)
- Complex Lesion
- Thrombectomy
- Lesion Preparation (pre-dilatation)
- Post-dilatation
- Use of Bailout Stent
- Total Number of Stents Implanted
- Post-procedure within stent after Post-dilatation
- Other concomitantly-used medical device

#### 3) Bifurcated Lesion (If applicable)

- Side Branch AHA Segment
- Bifurcation Lesion Type
- Technique Used
- Kissing Balloon



14-306 Version 1.0 

# 4) Lesion Visual Assessment (Pre and Post Procedure)

Angiographic corelab analysis data will be adopted when it is applicable.

- Lesion Length
- Reference Vessel Diameter
- %DS
- TIMI Flow

# 5) Stent Information

- Stent information must be recorded per lesion
  - Length and Diameter
  - o Deployment Pressure
  - o Successful Deployment
  - o Deployed Vessel (main vessel or side branch)

#### 5.3 Post Procedure Information

### 1) Post-Procedure ECG

#### 2) Post-Procedure

- Cardiac Enzyme
  - o CK
  - o CK-MB (If MI is suspected then must be measured per site standard practice)

#### 5.4 Post-Procedure (Maintenance) Antiplatelet

- Type
- Start Date
- Daily Dose
- Termination or Continuation

# 5.5 8 Months Follow-up

# 1) General Information

- Contact Method
- Contact Date
- Reportable adverse event since the last follow-up
- Change or termination of antiplatelet therapy
- Device Deficiency
- Follow-up Angiogram
- Ischemic Symptoms
- Revascularization

#### 2) Angiographic Information

Angiographic corelab analysis data will be adopted when it is applicable.

- Lesion Length (if restenosis exist)
- Reference Vessel Diameter
- %DS

# 5.6 1~5 Years Follow-up (Every Year)

- Contact Method
- Contact Date
- Reportable adverse event since the last follow-up
- Change or termination of antiplatelet therapy
- Device Deficiency

# 5.7 Unscheduled Visit (Reportable AE related)

Complete AE form(s) if a patient visits the hospital with reportable adverse event(s).

#### 5.8 Device Deficiency

- Date of deficiency
- Type of deficiency
- Did the device deficiency result in an adverse event?
- Description of deficiency/comment
- Product details (lot, serial numbers, etc.)



14-306 Version 1.0 

### 5.9 Adverse Event (Reportable Event)

Record the following adverse events (including procedural complications) and their details.

- All Coronary artery related adverse events
  - o Ischemic symptoms, evidences, including test results
  - o Diagnostic angiogram
  - o Revascularization
- All serious adverse events\*
- All events for which relationship to XIENCE Xpedition 2.25mm stent cannot be ruled out
- All other adverse events related to taking antiplatelet medication(s)
- \* Serious adverse event: death, life-threatening, hospitalization (initial or prolonged), disability or permanent damage, congenital anomaly/birth defect, other serious (investigator's judgment).

Evaluate and record relationship of the above adverse events to the Device, procedure, and antiplatelet therapy, as well as the outcome of each event. If the event is an SAE, record the reason for considering the event as an SAE.

#### 6. EVALUATION ITEMS

#### **6.1** Important Evaluation Items

Important evaluation items in this PMS are;

- 1) Stent Thrombosis
- 2) Adverse events caused by Anti-platelet Medications
- 3) Longitudinal stent deformation

#### **6.2** Other Evaluation Items

Other evaluation items will be per standard drug eluting studies.

#### 7. DATA ANALYSIS

# 7.1 Angiographic Core-Lab

Angiographic data at the index procedure and 8 months follow-up will be analyzed by Core-lab for lesion characteristics and quantitative coronary angiography (QCA) analysis.

Core-lab: KIC Co., Ltd Core-lab Department 34-15 Yanagi-cho Kanazawa-ku Yokohama city



14-306 Version 1.0 

# 7.2 Independent Review of Adverse Events

Objective review of adverse events (Stent Thrombosis, Cardiac Death, Myocardial Infarction, and TLR/TVR) will be conducted by a third party (medical professional) up to 3 years post index procedure. These events will be reviewed based on ARC definition. QCA results from angiographic core-lab will be provided to the reviewer as necessary.

#### 7.3 Analysis of Results

Collected data will be analyzed and Annual Report will be submitted according to "Survey Report on new medical device usage" (Japan Pharmaceutical and Food Safety Bureau Notice 1224, no. 4, dated December 24, 2010). Subgroup analyses will be conducted as necessary to evaluate safety and efficacy of the device, and included in the resubmission report.

The XIENCE Xpedition 2.25 mm stent is composed of the stent identical to the stent of the XIENCE PRIME SV Stent approved on March 7, 2013. Therefore, the data collected from the PMS will be pooled with data collected from the ongoing XIENCE PRIME SV PMS for analysis.